CLINICAL TRIAL: NCT01771185
Title: Metabolic Effects of Duodenal-jejunal Bypass Surgery in Non Morbidly Obese Subjects With Type 2 Diabetes
Brief Title: Metabolic Effects of Gastrointestinal Surgery in T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Cohen, Clinical Professor of Surgery, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUUSP001
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; metabolic surgery; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Metformin; Gliclazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best medical treatment (Active Comparator): Metformin 2 g/day; gliclazide 30 mg
  Interventions: Drug: Best medical treatment (Metformin ; gliclazide)
- Duodenal jejunal bypass plus sleeve gastrectomy (Active Comparator): Duodenal jejunal bypass plus sleeve gastrectomy is a metabolic surgical procedure
  Interventions: Procedure: Duodenal jejunal bypass plus sleeve gastrectomy

INTERVENTIONS:
Procedure: Duodenal jejunal bypass plus sleeve gastrectomy — Metabolic Surgery Duodenal jejunal bypass plus sleeve gastrectomy
  Arms: Duodenal jejunal bypass plus sleeve gastrectomy
Drug: Best medical treatment (Metformin ; gliclazide) — Metformin 2 g/day; gliclazide 30 mg
  Arms: Best medical treatment

SUMMARY:
Gastric bypass surgery resolves type 2 diabetes mellitus (T2DM) without the need for diabetes therapy in ~80% of patients. Moreover, improvement in insulin sensitivity and glucose homeostasis occurs within days after surgery before significant weight loss is achieved. This observation has led to the notion that bypassing the upper gastrointestinal (GI) tract has specific therapeutic effects on insulin action and glucose metabolism. In fact, both surgical and endoscopic procedures that bypass the upper GI tract are currently being studied in human subjects. Recently, a new surgical technique, duodenal-jejunal bypass surgery (DJBS), has been developed specifically to treat T2DM. Data from preliminary studies have shown that DJBS results in glycemic control in 87% of overweight and obese patients with T2DM.These subjects will undergo metabolic studies at the University Hospital in Sao Paulo before and after their surgical procedure. Washington University investigators will: 1) provide technical support and guidance to the physicians performing the studies in Brazil, 2) process and analyze blood samples obtained from the study at the Washington University Center for Human Nutrition, and 3) be involved in analyzing the data and writing the final manuscripts. The effects of DJBS on the following clinical and metabolic parameters will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled diabetes ( A1c>8%)
* Less than 10 years of history
* Not taking insulin
* Ages between 20 and 65 years old
* BMI between 26-34

Exclusion Criteria:

* previous abdominal surgery
* LADA
* Using insulin

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Hb A1a | 24 mo
  Primary endpoints- glycemic control

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure control | 24 mo
fasting glycemic control | 24 months
Lipidic control | 24 months